CLINICAL TRIAL: NCT01368614
Title: Randomized Controlled Trial Evaluating the Feasibility of AVAPS-AE vs. CPAP vs.Bilevel Pressure Support Ventilation in Obesity Hypoventilation Syndrome
Brief Title: AVAPS-AE Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRC-1006-AVAPS-AE-MS
Record Dates: First submitted 2011-05-23; First posted 2011-06-08 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Obesity Hypoventilation Syndrome
Keywords: OHS
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- AVAPS-AE (Experimental): AVAPS-AE Mode of ventilation
  Interventions: Device: AVAPS-AE Mode of Therapy
- Respironics OmniLab Advanced BiPAP S mode (Active Comparator): OmniLab Advanced BiPAP S Mode of ventilation
  Interventions: Device: Respironics OnmiLab BiPAP S mode
- Respironics OmniLab Advanced CPAP mode (Active Comparator): OmniLab Advanced CPAP Mode of ventilation
  Interventions: Device: Respironics OmniLab Advanced CPAP mode

INTERVENTIONS:
Device: AVAPS-AE Mode of Therapy — AVAPS-AE mode is the experimental mode of therapy in this study that includes a combination of already cleared therapy attributes.
  Arms: AVAPS-AE
Device: Respironics OnmiLab BiPAP S mode — Currently cleared Non-Invasive Ventilation (NIV) therapy modality
  Arms: Respironics OmniLab Advanced BiPAP S mode
Device: Respironics OmniLab Advanced CPAP mode — Currently cleared NIV therapy modality
  Arms: Respironics OmniLab Advanced CPAP mode

SUMMARY:
The purpose of this study is to evaluate the feasibility of using of the Average Volume Assured Pressure Support (AVAPS-AE) mode versus Continuous Positive Airway Pressure (CPAP) and bilevel pressure support ventilation (PSV) modes of ventilation in patients diagnosed with Obesity Hypoventilation syndrome (OHS).

The investigators believe the use of the AVAPS-AE mode of ventilation after 6 weeks will yield daytime gas exchange values which are equivalent or no worse when compared to using CPAP and bilevel PSV modes of ventilation in the OHS population.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age; less than or equal to 70 years of age
* Diagnosis of Obesity Hypoventilation Syndrome via a diagnostic sleep study in the past 3 months but have not initiated therapy

  * BMI greater than or equal to 30 kg/m2
  * Daytime PaCO2 greater than or equal to 45 mmHg
  * Apnea Hypopnea index (AHI) > 5
* Daytime pH > 7.35
* Forced Expiratory Volume at 1 second / forced vital capacity (FEV1/FVC) > 70%

Exclusion Criteria:

* Acutely ill, medically complicated or who are medically stable, or as otherwise determined by the investigator
* Respiratory alkalosis (pH > 7.45), per investigator discretion
* Emergency admissions on chronic respiratory failure
* Hospitalization for respiratory exacerbation < 6 weeks prior to screening visit
* Participants in whom PAP therapy is otherwise medically contraindicated
* Impaired upper airway function. For example, obstruction due to infections(laryngitis, epiglottis), craniofacial malformations, tumors, uvulopalatopharyngoplasty, presence of tracheostomy, or bilateral vocal cord palsy that does not allow tolerance of Non-invasive positive pressure ventilation (NPPV)
* Facial trauma, burns, surgery or anatomical abnormalities interfering with mask fit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-09-12 (Actual); Primary Completion 2013-05-30 (Actual); Study Completion 2013-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Parthasarathy, MD, Principal Investigator — Southern Arizona VA Healthcare; Babak Mokhlesi, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Arizona School of Medicine, Tucson, Arizona
  - University of Chicago, Chicago, Illinois

REFERENCES:
- [Derived] Lastra AC, Masa JF, Mokhlesi B. CPAP titration failure is not equivalent to long-term CPAP treatment failure in patients with obesity hypoventilation syndrome: a case series. J Clin Sleep Med. 2020 Nov 15;16(11):1975-1981. doi: 10.5664/jcsm.8712. PMID 32713421
- [Derived] Bhattacharjee R, Khalyfa A, Khalyfa AA, Mokhlesi B, Kheirandish-Gozal L, Almendros I, Peris E, Malhotra A, Gozal D. Exosomal Cargo Properties, Endothelial Function and Treatment of Obesity Hypoventilation Syndrome: A Proof of Concept Study. J Clin Sleep Med. 2018 May 15;14(5):797-807. doi: 10.5664/jcsm.7110. PMID 29734990

RESULTS

PARTICIPANT FLOW:
Groups:
- Screening Period: All study participants that were screened and signed consent.
- AVAPS-AE: AVAPS-AE mode is the experimental mode of therapy in this study that includes a combination of already cleared therapy attributes.
- Respironics OmniLab Advanced BiPAP S Mode: Non-Invasive Ventilation (NIV) therapy modality in the OmniLab Advanced BiPAP.
- Respironics OmniLab Advanced CPAP Mode: Non-Invasive Ventilation (NIV) therapy modality in the Respironics OmniLab Advanced CPAP
Period: Screening Period
Arm/Group | Screening Period | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Started | 90 | 0 | 0 | 0
Completed | 32 | 0 | 0 | 0
Not Completed | 58 | 0 | 0 | 0
Not completed — Screen Failure | 58 | 0 | 0 | 0
Period: Study Period
Arm/Group | Screening Period | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Started | 0 | 11 | 10 | 11
Completed | 0 | 10 | 8 | 8
Not Completed | 0 | 1 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants that signed the consent form are considered for the baseline demographics
Groups:
- All Study Participants: All study participants that signed the consent are included in the baseline characteristics to due the high screen failure rate and large number of participants that discontinued the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 41
  White | 33
  More than one race | 0
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 90
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 49.3 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Daytime Partial Pressure of Carbon Dioxide in Arterial Blood (PaCO2)
Description: Daytime PaCO2 measurements will be assessed for all randomized patients to each mode of ventilation therapy (AVAPS-AE, bilevel PSV, CPAP) after 6 weeks.
Time Frame: Screening & 6 weeks
Population: 6 participants withdrew from the study and therefore did not provide values at week 6.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Respironics OmniLab Advanced BiPAP S Mode: OmniLab Advanced BiPAP S Mode of ventilation
  Respironics OnmiLab BiPAP S mode: Currently cleared NIV therapy modality
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 11 | 10 | 11
mmHg
  Screening | 47.1 (2.5) | 51.8 (8.0) | 50.7 (4.7)
  Week 6: number analyzed (Participants) | 10 | 8 | 8
  Week 6 | 40.7 (3.7) | 47.4 (8.9) | 40.8 (5.8)

2. Secondary Outcome: Daytime Partial Pressure of Oxygen in Arterial Blood(Pa02)
Description: Daytime Pa02 measurements will be assessed for all randomized patients to each mode of ventilation therapy (AVAPS-AE, bilevel PSV, CPAP) after 6 weeks.
Time Frame: Screening & 6 weeks
Population: 6 participants withdrew from the study and therefore did not provide values at week 6.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 11 | 10 | 11
mmHg
  Screening | 62.8 (5.8) | 56.9 (10.7) | 62.6 (9.8)
  Week 6: number analyzed (Participants) | 10 | 8 | 8
  Week 6 | 65.0 (4.5) | 58.7 (14.7) | 66.2 (5.9)

3. Secondary Outcome: Apnea Hypopnea Index (AHI)
Description: The AHI is the number of apneas and hypopneas per hour of sleep. It will be evaluated during the screening sleep study and the 6 week follow up sleep study. AHI less than 5 is considered normal. For an Apnea-Hypopnea Index (or AHI) from 5 to 15 denotes mild sleep apnea. Fifteen to 30 is moderate, while a greater than 30 AHI is considered severe.
Time Frame: Screening & 6 weeks
Population: 6 participants withdrew from the study and therefore did not provide values at week 6.
  1 Participant did not have scorable data from the baseline PSG to calculate this measure.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 11 | 10 | 10
events per hour
  Screening | 84.5 (37.9) | 67.7 (23.9) | 85.4 (33.5)
  Titration | 16.1 (11.6) | 22.4 (11.1) | 30.1 (23.6)
  Week 6: number analyzed (Participants) | 10 | 8 | 8
  Week 6 | 15.5 (11.8) | 12.4 (14.8) | 7.4 (7.9)

4. Secondary Outcome: Epworth Sleepiness Scale
Description: Epworth Sleepiness scale is a measure of daytime sleepiness. It is a series of 8 questions answered on a scale of 0 to 3, 0 being no chance of dozing and 3 being a high chance of dozing. The range of the scale is 0 to 24. The higher the total score, the higher the chance of falling asleep.
Time Frame: Screening & 6 weeks
Population: 6 participants withdrew from the study and therefore did not provide values at week 6.
  1 participant did not complete the ESS at the end of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 11 | 10 | 11
units on a scale
  Screening | 14.9 (4.8) | 12.0 (5.2) | 11.5 (6.1)
  Week 6: number analyzed (Participants) | 9 | 8 | 8
  Week 6 | 9.8 (5.8) | 8.1 (6.1) | 5.9 (5.0)

5. Secondary Outcome: Severe Respiratory Insufficiency Questionnaire (SRIQ)
Description: The SRIQ is a 49 question survey. This survey asks questions about the past week. It is answered on a scale of -2 to 2 and converted to 1 to 5, 1 is completely untrue and 5 is always true. The questionnaire is broken down into 7 sections when scoring: respiratory complaints, physical functioning, attendant systems and sleep, social relationships, anxiety, psychological well-being and social functioning. Once each scale score is calculated. The average score can be calculated by taking the mean of the subscales. This process of transformation produces a score between 0 and 100 with higher values indicating a better health-related quality of life according to content of the scale.
Time Frame: Screening & 6 weeks
Population: 6 participants withdrew from the study and therefore did not provide values at week 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 11 | 10 | 11
units on a scale
  Screening | 52.0 (14.5) | 53.4 (14.5) | 60.0 (16.1)
  Week 6: number analyzed (Participants) | 10 | 8 | 8
  Week 6 | 61.0 (13.5) | 64.8 (18.4) | 69.7 (13.4)

6. Secondary Outcome: Ventilator Adherence - Average Hours
Description: The average number of hours ventilator was used per each day used.
Time Frame: 6 weeks
Population: 6 participants withdrew from the study and therefore did not provide values at week 6.
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 10 | 8 | 8
Hours per day | 4.8 (0.9) | 5.2 (1.7) | 6.6 (0.4)

7. Secondary Outcome: Ventilator Adherence - Days Used
Description: Average number of days used per week
Time Frame: 6 weeks
Population: 6 participants withdrew from the study and therefore did not provide values at week 6.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 10 | 8 | 8
days per week | 5.3 (0.9) | 5.3 (1.5) | 6.9 (0.5)

8. Secondary Outcome: Actigraphy
Description: Actigraphy is a method of measuring activity and sleep which is achieved by wearing a small watch-like device for an extended period of time. The data is intended to provide an objective measure of physical activity and sleep / week patterns during pre / post sleep studies and throughout the 6 weeks of home use.
Time Frame: Screening & 6 weeks
Population: Participants were asked to wear an actiwatch to measure actigraphy. Actigraphy was reviewed as part of the study however a detailed analysis was not conducted because the data was to variable.
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Room Air Sp02 Assessment Via Pulse Oximetry
Description: Oxygen saturation measurements as determined by pulse oximetry
Time Frame: Screening & 6 weeks
Population: 6 participants withdrew from the study and therefore did not provide values at week 6.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation (SpO2)
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 11 | 10 | 11
percentage of oxygen saturation (SpO2)
  Screening | 92.5 (3.4) | 90.6 (4.1) | 92.9 (2.5)
  Week 6: number analyzed (Participants) | 10 | 8 | 8
  Week 6 | 94.6 (2.0) | 90.1 (7.2) | 94.1 (2.5)

10. Secondary Outcome: Nocturnal Transcutaneous Capnography (TcC02)
Description: Nocturnal Transcutaneous Capnography is a non-invasive monitoring tool to measure ventilation over the night.
  .
Time Frame: Screening & 6 weeks
Population: This measure was not a standard practice of the sleep scoring company and was not done.
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Duration, Efficiency and Quality of Sleep and Sleepiness (Derived From Sleep Study) - Duration
Description: Duration, efficiency and quality of sleepiness are measured by a number of different parameters. Total sleep time in each stage provides the average amount of time a participant was in that stage of sleep. This includes Stage 1, Stage 2, Stage 3/4, and Rapid Eye Movement (REM) sleep.
Time Frame: Screening & 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of time spent in that stage
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 11 | 10 | 10
percentage of time spent in that stage
  Total Sleep Time Stage 1- Screening | 28.4 (19.5) | 24.6 (26.6) | 18.9 (15.6)
  Total Sleep Time Stage 1- 6 weeks: number analyzed (Participants) | 10 | 8 | 8
  Total Sleep Time Stage 1- 6 weeks | 10.0 (6.8) | 13.1 (10.3) | 10.1 (7.3)
  Total Sleep Time Stage 2- Screening | 50.8 (15.8) | 59.1 (22.4) | 64.8 (15.8)
  Total Sleep Time Stage 2-6 weeks: number analyzed (Participants) | 10 | 8 | 8
  Total Sleep Time Stage 2-6 weeks | 59.2 (15.1) | 52.4 (14.3) | 53.2 (15.4)
  Total Sleep Time Stage 3/4 - Screening | 8.5 (13.7) | 8.1 (11.7) | 7.8 (8.4)
  Total Sleep Time Stagev3/4-6 weeks: number analyzed (Participants) | 10 | 8 | 8
  Total Sleep Time Stagev3/4-6 weeks | 12.5 (13.2) | 14.0 (10.9) | 16.6 (15.8)
  Total Sleep Time Stage REM- Screening | 13.5 (7.4) | 8.2 (10.1) | 8.5 (5.1)
  Total Sleep Time Stage REM-6 weeks: number analyzed (Participants) | 10 | 8 | 8
  Total Sleep Time Stage REM-6 weeks | 18.3 (8.9) | 20.4 (9.1) | 20.1 (7.5)

12. Secondary Outcome: Duration and Quality of Sleep and Sleepiness (Derived From Sleep Study) - Sleep Efficiency
Description: Duration, efficiency and quality of sleepiness are measured by a number of different parameters. Sleep efficiency is measured by the total time a participant is spent asleep.
Time Frame: Screening & 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of time spent in that stage
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 11 | 10 | 10
percentage of time spent in that stage
  Sleep Efficiency - Screening | 74.4 (14.9) | 64.5 (14.9) | 74.6 (18.9)
  Sleep Efficiency - 6 weeks: number analyzed (Participants) | 10 | 8 | 8
  Sleep Efficiency - 6 weeks | 86.8 (8.4) | 71.4 (17.1) | 74.4 (23.8)

13. Secondary Outcome: Duration, Efficiency and Quality of Sleep and Sleepiness (Derived From Sleep Study)- Arousal and Awakening Indices
Description: The arousal index is measured by the average number of arousals or awakenings a participant has over an hour of sleep.
Time Frame: Screening & 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: arousals per hour
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 11 | 10 | 10
arousals per hour
  Screening | 68.2 (31.2) | 66.0 (20.9) | 71.4 (27.1)
  6 weeks: number analyzed (Participants) | 10 | 8 | 8
  6 weeks | 19.4 (9.3) | 23.0 (10.9) | 21.3 (10.1)

14. Secondary Outcome: Duration, Efficiency and Quality of Sleep and Sleepiness (Derived From Sleep Study)- Nocturnal O2 Saturation
Description: Measurement of overnight oxygen saturation as measured by percentage of oxygen saturation (SpO2)
Time Frame: Screening & 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation (SpO2)
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 11 | 10 | 10
percentage of oxygen saturation (SpO2)
  Screening | 84.2 (6.0) | 81.6 (7.5) | 81.1 (8.5)
  6 weeks: number analyzed (Participants) | 10 | 8 | 8
  6 weeks | 92.7 (2.5) | 93.3 (2.9) | 94.5 (1.4)

15. Secondary Outcome: Reaction Time (Psychomotor Vigilance Test-PVT)
Description: To measure trends of vigilance between the baseline screening assessment and the 6 week follow up visit comparing the three Arms/Groups. This measured how quickly participants reacted to visual stimulus. Reaction time is the latency at which the participant reacts to a visual stimulus > 100 ms.
Time Frame: Screening & 6 weeks
Population: 1. participant from the AVAPS-AE Arm/Group did not complete the baseline screening PVT.
  2. participants from the Omnilab Advanced BIPAP Arm/Group did not complete the 6 week follow up PVT.
  3. participants from the Omnilab Advanced CPAP Arm/Group did not complete the 6 week follow up PVT.
Measure: Median (Standard Deviation); unit: milliseconds
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 9 | 8 | 8
milliseconds
  Screening: number analyzed (Participants) | 8 | 8 | 8
  Screening | 3987.13 (8441.71) | 4752.75 (11435.85) | 4523.25 (10820.36)
  6 weeks: number analyzed (Participants) | 9 | 6 | 5
  6 weeks | 2978.89 (7133.21) | 5681.83 (12593.01) | 6705.20 (13840.41)

16. Secondary Outcome: Number of Participants With Need for Continued Oxygen Supplementation
Description: Some users enrolled into the study required supplemental oxygen at different times during the day: at rest, during exertion and at night. The need for supplemental oxygen was compared at baseline and at 6 weeks.
Time Frame: Screening & 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
Number analyzed (Participants) | 11 | 10 | 11
Participants
  At Rest- Screening | 1 | 4 | 0
  At Rest-6 weeks | 0 | 2 | 1
  At Sleep- Screening | 2 | 4 | 0
  At Sleep- 6 weeks | 0 | 2 | 1
  At Exertion- Screening | 0 | 1 | 0
  At Exertion- 6 weeks | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: All Adverse Events experienced over 6 weeks were collected.
Arm/Group | AVAPS-AE | Respironics OmniLab Advanced BiPAP S Mode | Respironics OmniLab Advanced CPAP Mode
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 2/11
Other Adverse Events (participants affected / at risk) | 1/11 | 0/10 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVAPS-AE (N=11) | Respironics OmniLab Advanced BiPAP S Mode (N=10) | Respironics OmniLab Advanced CPAP Mode (N=11)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fournier's Gangrene (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVAPS-AE (N=11) | Respironics OmniLab Advanced BiPAP S Mode (N=10) | Respironics OmniLab Advanced CPAP Mode (N=11)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No